CLINICAL TRIAL: NCT05684276
Title: Phase II Clinical Trial of Neo-adjuvant Chemo/Immunotherapy Followed by Adjuvant Treatment Depending on the Resection Status for the Treatment of NSCLC Patients Diagnosed With Pancoast Tumor. A Multicenter Exploratory Study
Brief Title: DUMAS: Neo-Adjuvant Immunotherapy for Pancoast Tumors
Acronym: DUMAS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fundación GECP (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GECP 22/02_DUMAS; 2022-003717-11 (EudraCT Number)
Record Dates: First submitted 2023-01-05; First posted 2023-01-13 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: NSCLC; Pancoast Tumor
Keywords: Neoadjuvant Treatment; Nivolumab
MeSH Terms: conditions — Pancoast Syndrome | interventions — Carboplatin; Paclitaxel; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Neodjuvant treatment + Adjuvant maintenance treatment (Experimental): Neodjuvant treatment:
  Nivolumab: 360 mg intravenous Q3W Paclitaxel: 200mg/m2 infusion over 3 hours Carboplatin: AUC6 at the end of the Paclitaxel infusion
  Neoadjuvant treatment will start within 1-3 days from enrollment. 3 cycles will be administered at 21-day (+/- 3 days) intervals (QW3) prior to surgery. Before surgery a tumor assessment will be done. Patients must leave the study if there is evidence of progression. Patients with stable disease or partial response may be considered for surgery.
  Surgery: Surgery must be done within the 3rd-4th week (+7 days) from day 21 cycle 3 of neoadjuvant treatment (day 42-49 after day 1 of cycle 3)
  Depending on surgery results the patient will receive:
  * Patients with degree of resection 'R0': Adjuvant treatment for 6 months with Nivolumab 480mg QW4
  * Patients with degree of resection 'R1' or 'R2': standard treatment according to local guidelines
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: Nivolumab

INTERVENTIONS:
Drug: Carboplatin — Structure: The cis-diamino (cyclobutane-1, 1 dicarboxylate) plating. Stability: 24 hours at ambient temperature in 5% glucose, sodium chloride and glucose 5% solution solution or physiologic saline. It is recommended not to dilute with chlorinated solutions for this could affect the carboplatin.
  Route of administration: Intravenous infusion. Guidelines of Carboplatin administration: According to the standard of ech center.
  Other Names: Paraplatin
Drug: Paclitaxel — Structure: A diterpene whose composition is: 5b, 20-epoxy-1, 2a, 4,7b, 10b, 13a-hexa-hydroxy-11-en 9 one 4,10-diacetate 2-benzoate 13-ester with (2R,3S)- N-benzoyl-3-phenylisoserine.
  Stability: Concentrations of 0.3-1.2 mg/ml in 5% dextrose or normal saline have demonstrated chemical and physical stability for more that 27 hours at ambient temperature (25ºC approximately). The intact vial must be stored between 15º and 25ºC.
  Guidelines on Paclitaxel administration: Paclitaxel must be administered by infusion over 3 hours in dextrose (D5W) or normal saline (NS). The concentration must not exceed 1.2 mg/ml.
  Other Names: Taxol
Drug: Nivolumab — Structure: Nivolumab is a soluble protein consisting of 4 polypeptide chains. Route of administration: Intravenous infusion. Product Description: Nivolumab (BMS-936558-01) Injection drug product is a sterile, non-pyrogenic, single-use, isotonic aqueous solution formulated in 10 mg/ml.
  Storage Conditions: It must be stored at 2 to 8 degrees Cº and protected from light and freezing.
  Guidelines: The administration of nivolumab infusion must be completed within 24 hours of preparation.The dose of Nivolumab for the adjuvant treatment is 360 mg administered as an intravenous infusion over 30 minutes every 3 weeks (+/-3 days) for 3 cycles.
  For the maintenance adjuvant treatment the dose is nivolumab 480 mg Q4W (+/-3 days) over 30 minutes for 6 months (6 cycles).
  Subjects should be carefully monitored during nivolumab administration to follow infusion reactions. Doses of nivolumab may be interrupted, delayed, or discontinued depending on how well the subject tolerates the treatment.
  Other Names: Opdivo

SUMMARY:
The goal of this clinical trial is to test the efficacy of induction treatment of immunotherapy and chemotherapy depending on the resection status for the treatment of non small cell lung cancer patients diagnosed with pancoast tumor.

The main objectives it aims to answer are:

* Complete resection rate after induction treatment with chemotherapy plus nivolumab
* Overall Survival and Progression Free Survival at 24 months

The sample size is 40 patients.

DETAILED DESCRIPTION:
This is an open-label, phase II, single-arm, multi-centre clinical trial.

The total sample size is 40 patients. The population to be included are previously untreated patients with histologically- or cytologically- documented NSCLC diagnosed with Pancoast tumor.

Patients will receive Nivolumab 360mg + Paclitaxel 200mg/m2 + Carboplatin AUC6 for 3 cycles every 21 days (+/- 3 days) as neoadjuvant treatment followed by surgery and 6 months of adjuvant treatment with Nivolumab 480 mg Q4W (+/- 3 days) if applicable and depending on surgery results. Patients that will not receive adjuvant treatment will start follow up phase after end of treatment visit. Follow up for all patients must be done for 2 years.

The primary objective is to evaluate the complete resection (R0) rate after induction treatment defined as the absence of residual tumor in patients treated with neoadjuvant chemo-immunotherapy.Secondary objectives and endpoint are Overall survival rate at 24 months and disease-free survival rate at 24 months.

Patient accrual is expected to be completed within 2 years excluding a run-in-period of 3 months. Treatment and follow-up are expected to extend the study duration to a total of 5 years. The study will end once survival follow-up has concluded.

ELIGIBILITY:
Inclusion Criteria:

* 1. Previously untreated patients with histologically- or cytologically- documented NSCLC diagnosed with Pancoast tumor according to 8th edition of the TNM (stages IIB, IIIA and T3N2 (IIIB) patients)
* 2. PET/CT including IV contrast (CT of diagnostic quality) will be performed at baseline (28 days +10 before enrollment) to rule out the presence of distant disease. Also, a brain CT-SCAN or brain MRI will be done at baseline
* 3. Positive mediastinal lymph nodes by PET-CT must be confirmed histologically. Mediastinal involvement may be considered without the need for histological confirmation when there is a mass of lymph nodes in which the margins cannot be distinguished
* 4. Measurable or evaluable disease (according to RECIST 1.1 criteria)
* 5. ECOG (Performance status) 0-2
* 6. Patients with a life expectancy of at least more than 12 weeks
* 7. Patients aged > 18 years and ≤ 75 years
* 8 Screening laboratory values must meet the study criteria and should be obtained within 14 days prior to enrollment
* 9. Correct lung function without bronchodilators, defined by forced expiratory volume in 1 second (FEV1) >40% of the predicted normal volume, and a pulmonary diffusing capacity for carbon monoxide (DLCO) >40% of the predicted normal value
* 10. All patients are notified of the investigational nature of this study and signed a written informed consent in accordance with institutional and national guidelines, including the Declaration of Helsinki prior to any trial-related intervention
* 11. Women of childbearing potential, including women who had their last menstrual period in the last 2 years, must have a negative serum or urine pregnancy test within 7 days before enrollment.
* 12. All sexually active men and women of childbearing potential must use an effective contraceptive method during the study treatment and for a period of at least 12 months following the last administration of trial drugs
* 13. Patient capable of proper therapeutic compliance and accessible for correct follow-up.

Exclusion Criteria:

* 1. Patients that receive previous treatment with antineoplastic drugs, chest radiotherapy, or previous surgery for lung cancer or for another reason
* 2. Pleural or pericardial effusion: Both will be considered indicative of metastatic disease unless proven otherwise. Those that, even being cytologically negative for malignancy, are exudates, will also be excluded. Patients with pleural effusion not visible on chest X-ray or too small to perform diagnostic puncture safely may be included.
* 3. Patients with a weight loss >10% in the 3 months prior to the study entry
* 4. All patients carrying activating mutations in the TK domain of EGFR or any variety of alterations in the ALK gene or ROS1 mutations.
* 5. Patients with active, known or suspected autoimmune disease. Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune thyroiditis only requiring hormone replacement or unexpected conditions of recurrence in the absence of an external trigger are allowed to be included.
* 6. Patients with symptomatic neuropathy > grade 1 according to the CTCAE v5.0 and that were not related to the tumor
* 7. Patients with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of enrollment. Inhaled or topical steroids, and adrenal replacement steroid doses > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
* 8. Patients with a history of interstitial lung disease cannot be included if they have symptomatic ILD (Grade 3-4) and/or poor lung function. In case of doubt please contact trial team.
* 9. Patients with other active malignancy requiring concurrent intervention and/or concurrent treatment with other investigational drugs or anticancer therapy
* 10. Patients with uncontrolled comorbidities that may affect the clinical trial compliance
* 11. Patients with previous malignancies (except non-melanoma skin cancers, and the following in situ cancers: bladder, gastric, colon, endometrial, cervical/dysplasia, melanoma, or breast) are excluded unless a complete remission was achieved at least 5 years prior to study entry and no additional therapy is required during the study period.
* 12. Any medical, mental, neurological or psychological condition which in the opinion of the investigator would not permit the patient to complete the study or understand the patient information sheet.
* 13. Patients in any psychological, familiar, sociological or geographical situation that may hinder compliance with the study protocol and/or the follow up
* 14. Patients who have had prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways
* 15. Patients with positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection
* 16. Patients with known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
* 17. Patients with know hypersensitivity to drugs with a structure similar to the study drug and/or history of allergy to study drug components excipients
* 18. Women who are pregnant or in the period of breastfeeding
* 19. Sexually active men and women of childbearing potential who are not willing to use an effective contraceptive method during the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2023-05-12 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Estimate progression-free survival (PFS) | From the date randomization until the date of last follow up, assessed up to 24 months
  The PFS is defined as the time from diagnosis to relapse, progression or death, whichever occurred first

SECONDARY OUTCOMES:
Overall survival | From the date of randomization until the date of last follow up, assessed up to 24 months
  The length of time from either the date of diagnosis or the start of the treatment that patients diagnosed with the disease are still alive.
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | From the subject's written consent to participate in the study through 100 days after the final administration of the drug
  It will be measured by the incidence of AE, SAE, immune-related AEs, deaths, and laboratory abnormalities. Adverse events will be graded according to CTCAE v5.0
Complete resection (R0) rate | From the date of completion of induction treatment until the date of last follow up, assessed up to 24 months
  Defined as the time between the date of randomization and the date of death

CONTACTS AND LOCATIONS:
Overall Officials: Mariano Provencio, MD, Study Chair — Fundación GECP President
Locations (29):
- Spain (29):
  - Hospital De Mataro, Mataró, Barcelona
  - Hospital Universitario Jerez De La Frontera, Jerez de la Frontera, Cádiz
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Hospital General Universitario de Elche, Alicante
  - Hospital Universitari Quiron Dexeus, Barcelona
  - Hospital Universitari Vall d' Hebron, Barcelona
  - Hospital Clínic De Barcelona, Barcelona
  - Hospital Parc Taulí, Barcelona
  - Hospital Universitario de Cruces, Bilbao
  - Hospital San Pedro De Alcántara, Cáceres
  - Hospital Josep Trueta, Girona
  - Hospital Universitario de Jaén, Jaén
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital 12 De Octubre, Madrid
  - Hospital Universitario la Paz, Madrid
  - Fundació Althaïa, Manresa
  - Hospital Universitario Regional de Málaga, Málaga
  - Hospital Son Espases, Palma de Mallorca
  - Hospital Universitario Salamanca, Salamanca
  - Hospital Universitario Virgen Del Rocio, Seville
  - Consorci Sanitari de Terrassa, Terrassa
  - Hospital Clínico de Valencia, Valencia
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Universitario Dr. Peset, Valencia
  - Hospital Universitario La Fe, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid
  - Complexo Hospitalario Universitario De Vigo, Vigo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Web page of the sponsor where users can find more information about Fundación GECP studies — http://www.gecp.org